CLINICAL TRIAL: NCT00310973
Title: HIV Prevention Within High-Risk Social Networks
Brief Title: HIV Prevention Within High-Risk Bulgarian and Hungarian Social Networks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kelly, Professor and Director, Center for AIDS Intervention Research, Medical College of Wisconsin
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH064410 (NIH); R01MH064410 (NIH); DAHBR 9A-ASPG
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: HIV Infections
Keywords: HIV; Prevention; Risk Behavior Reduction; Roma; Bulgaria; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Social Network Intervention

SUMMARY:
This study will evaluate the effectiveness of peer-led HIV/sexually transmitted disease (STD)risk reduction educational counseling in reducing HIV risk behavior among the social networks of young men who have sex with men and Roma men and women in Bulgaria and Hungary.

DETAILED DESCRIPTION:
HIV is spreading more rapidly in Eastern Europe than anywhere else in the world. Bulgaria and Hungary are still in the early stages of the crisis. However, without efforts to prevent the spread of HIV and AIDS, both countries are likely to fall victim to the HIV/AIDS growth curve that has already affected the rest of Eastern Europe. Bulgarian and Hungarian young men who have sex with men (YMSM) and Roma men and women are at the greatest risk for HIV infection. In both countries, HIV is spread primarily through sexual transmission. Prevention efforts that are undertaken now could help these countries avoid an explosive HIV/AIDS epidemic. YMSM and Roma men in Bulgaria and Hungary are more likely to trust HIV/AIDS information received from someone they know than from an official statement. Therefore, entire social networks will be recruited for this study and the leader of each network will be responsible for delivering the prevention information to his or her peers. This study will evaluate the effectiveness of peer-led HIV/STD risk reduction educational counseling in reducing HIV risk behavior among the social networks of YMSM and Roma men and women in Bulgaria and Hungary.

This study will recruit 40 YMSM and 40 Roma high-risk social networks. Each network will be randomly assigned to receive either standard HIV/AIDS risk reduction or the intervention. Networks assigned to receive the intervention will be assessed sociometrically to determine the 'social influence' leaders of each group. The leaders will then attend a 9-session program over the course of 3 months that will train them to deliver theory-based risk-reduction messages and peer-counseling to their respective social networks. The messages will focus on promoting safer sex knowledge, attitudes, intentions, perceived norms, and self-efficacy. All participants will be offered STD testing and their HIV-risk behavior will be assessed at Months 3 and 12. Participants assigned to receive the standard HIV/AIDS risk reduction will then receive the network intervention for an additional 12 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 50% of social network members complete baseline assessments
* At least 50% of assessed members of a social network report unprotected vaginal or anal intercourse outside of a mutually monogamous relationship in the 6 months prior to study entry

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2003-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Reductions in the prevalence and frequency of unprotected vaginal or anal intercourse | Months 3 and 12 post intervention

SECONDARY OUTCOMES:
Lower incidence of sexually transmitted diseases | Months 3 and 12 post intervention
Change in AIDS-related scales | Months 3 and 12 post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin; Yuri A. Amirkhanian, PhD, Study Director — Medical College of Wisconsin
Locations (3):
- Health and Social Development Foundation, Sofia, Bulgaria
- Institute of Sociology, Hungarian Academy of Sciences, Budapest, Hungary
- Botkin Hospital for Infectious Diseases, Saint Petersburg, Russia

REFERENCES:
- [Result] Kabakchieva E, Vassileva S, Kelly JA, Amirkhanian YA, DiFranceisco WJ, McAuliffe TL, Antonova R, Mihaylova M, Vassilev B, Khoursine R, Petrova E. HIV risk behavior patterns, predictors, and sexually transmitted disease prevalence in the social networks of young Roma (Gypsy) men in Sofia, Bulgaria. Sex Transm Dis. 2006 Aug;33(8):485-90. doi: 10.1097/01.olq.0000204533.20324.56. PMID 16641823
- [Result] Amirkhanian YA, Kelly JA, Kabakchieva E, Kirsanova AV, Vassileva S, Takacs J, DiFranceisco WJ, McAuliffe TL, Khoursine RA, Mocsonaki L. A randomized social network HIV prevention trial with young men who have sex with men in Russia and Bulgaria. AIDS. 2005 Nov 4;19(16):1897-905. doi: 10.1097/01.aids.0000189867.74806.fb. PMID 16227798
- [Result] Takacs J, Amirkhanian YA, Kelly JA, Kirsanova AV, Khoursine RA, Mocsonaki L. "Condoms are reliable but I am not": A qualitative analysis of AIDS-related beliefs and attitudes of young heterosexual adults in Budapest, Hungary, and St. Petersburg, Russia. Cent Eur J Public Health. 2006 Jun;14(2):59-66. doi: 10.21101/cejph.a3373. PMID 16830606
- [Result] Amirkhanian YA, Kelly JA, Kirsanova AV, DiFranceisco W, Khoursine RA, Semenov AV, Rozmanova VN. HIV risk behaviour patterns, predictors, and sexually transmitted disease prevalence in the social networks of young men who have sex with men in St Petersburg, Russia. Int J STD AIDS. 2006 Jan;17(1):50-6. doi: 10.1258/095646206775220504. PMID 16409680
- [Result] Amirkhanian YA, Kelly JA, Kabakchieva E, McAuliffe TL, Vassileva S. Evaluation of a social network HIV prevention intervention program for young men who have sex with men in Russia and Bulgaria. AIDS Educ Prev. 2003 Jun;15(3):205-20. doi: 10.1521/aeap.15.4.205.23832. PMID 12866833
- [Result] Kelly JA, Amirkhanian YA, Kabakchieva E, Csepe P, Seal DW, Antonova R, Mihaylov A, Gyukits G. Gender roles and HIV sexual risk vulnerability of Roma (Gypsies) men and women in Bulgaria and Hungary: an ethnographic study. AIDS Care. 2004 Feb;16(2):231-45. doi: 10.1080/09540120410001641075. PMID 14676028
- [Result] Amirkhanian YA, Kelly JA, McAuliffe TL. Identifying, recruiting, and assessing social networks at high risk for HIV/AIDS: methodology, practice, and a case study in St Petersburg, Russia. AIDS Care. 2005 Jan;17(1):58-75. doi: 10.1080/09540120412331305133. PMID 15832834
- [Derived] Kelly JA, Amirkhanian YA, Kabakchieva E, Vassileva S, Vassilev B, McAuliffe TL, DiFranceisco WJ, Antonova R, Petrova E, Khoursine RA, Dimitrov B. Prevention of HIV and sexually transmitted diseases in high risk social networks of young Roma (Gypsy) men in Bulgaria: randomised controlled trial. BMJ. 2006 Nov 25;333(7578):1098. doi: 10.1136/bmj.38992.478299.55. Epub 2006 Oct 13. PMID 17040924